CLINICAL TRIAL: NCT06329583
Title: Establishing Pressures at the Esophagogastric Junction During Diaphragmatic Breathing Using High-resolution Esophageal Manometry
Brief Title: Establishing Pressures at the EGJ During Diaphragmatic Breathing Using High-resolution Esophageal Manometry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andree H. Koop, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-012635
Record Dates: First submitted 2024-03-14; First posted 2024-03-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Gastroesophageal Reflux; Dysphagia; Esophageal Motility Disorders
MeSH Terms: conditions — Gastroesophageal Reflux; Deglutition Disorders; Esophageal Motility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diaphragmatic breathing protocol (Other): All patients will undergo the diaphragmatic breathing protocol with high-resolution esophageal manometry.
  Interventions: Diagnostic Test: diaphragmatic breathing

INTERVENTIONS:
Diagnostic Test: diaphragmatic breathing — Different positions and techniques for diaphragmatic breathing

SUMMARY:
The goal of this study is to determine which position, maneuvers or combination thereof generates the highest pressure at the EGJ as assessed by high-resolution esophageal manometry and thus greater or more robust contraction of the diaphragm.

DETAILED DESCRIPTION:
This is a prospective, single-center study of adult (age ≥18 years) participants undergoing high-resolution esophageal manometry to assess the optimal method of diaphragmatic breathing. Included patients will complete two validated surveys, the Brief Esophageal Dysphagia Questionnaire (BEDQ) and the Gastroesophageal Reflux Disease Questionnaire (GERDQ). Patients will then undergo a standard protocol of supine and upright swallows with high-resolution manometry analyzed according to the Chicago Classification v4.0. After completion of the standard manometry protocol, participants will then perform a protocol assessing different techniques and positions for diaphragmatic breathing.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing high-resolution esophageal manometry

Exclusion Criteria:

* prior esophageal or gastric surgery
* chest tube
* major concomitant illness
* sinus disease precluding manometry placement
* history of heavy alcohol or tobacco use
* poor comprehension and/or fluency of English language
* inability or unwillingness of individual to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pressure at the esophagogastric junction | Measured for each participant during high-resolution esophageal manometry. Data will be collected over the enrollment period of one year.
  Measurement of EGJ- contractile integral and diaphragmatic pressure with each exercise/instruction

CONTACTS AND LOCATIONS:
Overall Officials: Andree Koop, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials